CLINICAL TRIAL: NCT02344394
Title: Prospective, Randomized Comparison of Hybrid Ablation and Pulmonary Vein Isolation Alone Versus Hybrid Ablation With Pulmonary Vein Isolation Plus Catheter Ablation for CFAE and Linear Lesions
Brief Title: Comparison of Hybrid Ablation and Pulmonary Vein Isolation Alone vs Hybrid Ablation With PVI Plus Catheter Ablation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients did not want to be randomized in hybrid ablation.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-52
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2018-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Anti-Arrhythmia Agents; Catheter Ablation; surgical hybrid ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid Ablation-cryoballoon alone (Other): This group receives the hybrid surgical ablation (epicardial-endocardial ablation) with epicardial ablation and endocardial ablation consisting of pulmonary vein isolation with no further catheter ablation. This will be achieved using the nContact and Medtronic cryoballoon
  Interventions: Device: Medtronic Cryoballoon; Device: nContact
- Hybrid ablation-cryoballoon plus RF (Other): This group receives the hybrid surgical ablation (epicardial-endocardial ablation) with epicardial ablation and endocardial ablation. Endocardial portion consists of pulmonary vein isolation using the cryoballoon with further catheter ablation, which may consist of ablation of complex fractionated electrograms and linear lesions. This will be achieved using the nContact and Medtronic Cryoballoon plus Thermocool Catheter.
  Interventions: Device: Medtronic Cryoballoon; Device: Thermocool Catheter; Device: nContact

INTERVENTIONS:
Device: Medtronic Cryoballoon — For endocardial pulmonary vein Isolation, an Arctic Front Advance Cardiac CryoAblation catheter (Medtronic, Mounds view, MN, USA) will be used.
Device: Thermocool Catheter — For mapping and ablation from endocardium a 3.5 mm irrigated tip catheter (Navistar Thermocool SmartTouch Unidirectional Navigation Catheter, Biosense Webster, Diamond Bar, CA, USA) will be used.
  Arms: Hybrid ablation-cryoballoon plus RF
Device: nContact — For Epicardial Ablation (the surgical portion of the Hybrid procedure), we will use the VisiTrax cardiac ablation device (nContact, Morrisville, NC, USA).

SUMMARY:
The overall objective of the study is to compare and assess the clinical outcomes of the standard of care hybrid ablation using epicardial ablation in conjunction with endocardial PVI alone versus epicardial ablation in conjunction with endocardial ablation using PVI with additional RF ablation in a randomized, prospective population of patients with persistent AF of at least 6 months duration. All devices that are used are being utilized under the approved labeling of the devices.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the leading causes of stroke and heart failure. It is also a major cause of hospitalizations and mortality (Stewart, Wattigney, and Wolf). Patients with atrial fibrillation (AF) who are intolerant to Class I and III antiarrhythmic drugs often require endocardial ablation, which can include pulmonary vein isolation (PVI) using radiofrequency (RF) catheter ablation or cryoballoon ablation (Medtronic, MN) and reported success rates vary (Calkins et al). In patients with persistent and long standing persistent AF success rates may not be as high (Akoum et al) and there is little data analyzing outcomes for patients in this population (Calkins et al). Using an epicardial-endocardial, or hybrid, approach Gehi et al describes a 66% 12 month arrythmia-free survival rate following the procedure, with 37% patients still on antiarrythmic drug therapy at 12 months. Furthermore, a paper by Anderson et al reports that the hybrid ablation results in lower costs and higher quality adjusted life years for patients with non-paroxysmal AF as reported by the studie's results of fewer repeat ablations and maintenance of sinus rhythm at 5 years. Conflicting reports exist on how much endocardial catheter ablation is needed for patients in persistent and long standing persistent AF. Verma et al reports results for patients in persistent AF having endocardial PVI compared to P VI plus additional linear lesions. Eighteen month success rates for these patients were 59% and 46% respectively.

Success of surgical hybrid ablation using epicardial ablation cocontaminent with endocardial PVI alone versus the hybrid approach using epicardial ablation with endocardial ablation consisting of PVI ablation and RF ablation has not been studied using a randomized, prospective approach.

If it is found that the PVI alone is as effective as PVI plus additional catheter ablation for patients receiving a hybrid ablation, it may reduce the need for extensive catheter ablation, thereby reducing the radiation exposure, procedure time, and radiofrequency ablation time.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years of age or older
* Left atrium < 6.0 em (Trans Thoracic Echo - TTE- parasternal4 chamber view performed within 6 months)
* History of AF for at least 6 months
* Failed or refractory to one AAD (class I and/or Ill)
* Documentation of persistent AF
* Provided written informed consent
* Be eligible for the hybrid procedure

Exclusion Criteria:

* Pregnant or planning to become pregnant during study
* Co-morbid medical conditions that limit one year life expectancy
* Previous cardiac surgery
* Previous abdominal surgery which will prevent epicardial access
* History of pericarditis
* Previous cerebrovascular accident (CVA), excluding fully resolved TIA
* Patients who have active infection or sepsis
* Patients with esophageal ulcers strictures and varices
* Patients with renal dysfunction who are not on dialysis (defined as GFR ::5 40)
* Patients who are contraindicated for anticoagulants such as heparin and coumadin
* Patients who are being treated for ventricular arrhythmias
* Patients who have had a previous left atrial catheter ablation for AF (does not include ablation for AFL or other supraventricular arrhythmias)
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment
* Not competent to legally represent him or herself (e.g., requires a guardian or caretaker as a legal representative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Success or failure in patient with persistent AF to be free of 1) AF/Atrial tachycardia(AT)/Atrial flutter(AFL) and 2) class I and Ill antiarrhythmic drugs (AAD) | 12 months
  The primary endpoint is success or failure in patients with persistent AF of at least 6 months duration to be AF/Atrial tachycardia (AT)/Atrial flutter (AFL) free and free of class I and III antiarrhythmic drugs (AAD) except for a previously failed or intolerant AAD in the same class following the 3 month blanking period through the 12 months post procedure follow-up visit. A failed AAD is defined as recurrence on that particular AAD.
  Crossover: After the three month blanking period, if the patient is in persistent AF, the patient may undergo DCCV and antiarrhythmic medication started. The follow up will start after this date.

SECONDARY OUTCOMES:
Success or failure in patient with persistent AF to achieve a >90% reduction in AF burden and freedom of class I and Ill antiarrhythmic drugs (AAD) | 12 months
  Success or failure in patient with persistent AF of at least 6 months duration to achieve a >90% reduction in AF burden and freedom of class I and III antiarrhythmic drugs (AAD) except for a previously failed or intolerant AAD in the same class following the 3 month blanking period through the 12 months post procedure follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jasbir S Sra, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, St. Luke's Medical Center, Milwaukee, Wisconsin, United States